CLINICAL TRIAL: NCT01314066
Title: Efficacy of Bevacizumab in Preventing Acute Respiratory Distress Syndrome (ARDS)
Acronym: VEGF-ARDS
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No funding
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: IRB Protocol #0907010498
Record Dates: First submitted 2010-07-28; First posted 2011-03-14 (Estimated); Last update posted 2016-05-03 (Estimated); Status verified 2016-04

CONDITIONS: Severe Sepsis; Acute Respiratory Distress Syndrome
MeSH Terms: conditions — Sepsis; Respiratory Distress Syndrome | interventions — Bevacizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Bevacizumab 5 mg/kg (Experimental): Receive drug solution as a single dose. Treatment will be given as 90 minute IV infusion.
  Interventions: Drug: Bevacizumab
- Bevacizumab at 10 mg/kg (Experimental): Receive drug solution as a single dose. Treatment will be given as 90 minute IV infusion.
  Interventions: Drug: Bevacizumab
- Placebo (Placebo Comparator): In addition to receiving the best standard supportive care for both diagnosis and treatment for individuals diagnosed with severe sepsis, they will receive an IV saline solution.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Bevacizumab — Patients receiving drug will receive it as a single dose. Treatment will be given as 90-minute IV infusion. The patient will either receive Bevacizumab at 5 mg/kg OR Bevacizumab at 10 mg/kg.
  Other Names: Avastin
  Arms: Bevacizumab 5 mg/kg; Bevacizumab at 10 mg/kg
Drug: Placebo — Patients assigned to placebo-control group will receive a single dose of saline solution as a 90 minute IV infusion
  Arms: Placebo

SUMMARY:
This study aims to test the effectiveness of a single intravenous (IV, through the vein) dose of the study drug, bevacizumab (Avastin), in preventing/reducing the development of Acute Respiratory Distress Syndrome (ARDS), in patients with severe sepsis, who are at high risk for developing ARDS. ARDS is a lung disease caused by a lung injury that leads to lung function impairment. The condition the patient has,severe sepsis, is a medical condition associated with an infection characterized as an immune system inflammatory response throughout your whole body that can lead to organ dysfunction, low blood pressure or insufficient blood flow to one or more of your organs.

DETAILED DESCRIPTION:
Acute respiratory distress syndrome (ARDS) is the most extreme form of acute lung injury (ALI) that results in a loss of lung function and structure. Vascular endothelial growth factor (VEGF), a protein critical for lung development that is found in the thin layer of liquid lining the inner surface of the lung air sacs, is believed to play a key role in the development of ARDS. During ARDS/ALI, VEGF markedly increases the permeability of the cells lining the inner surface of blood vessels in the lungs, which leads to an accumulation of fluid in the lungs (pulmonary edema), a characteristic of ARDS/ALI. Thus, anti-VEGF therapies offer a unique approach to treat this potentially fatal disorder. Bevacizumab (Avastin ®), an anti-VEGF medication, has been shown to be effective in inhibiting pulmonary edema caused by VEGF over-expression in an animal model.

This study will establish the usefulness and effectiveness of a singe dose of Bevacizumab administered intravenously (through the vein) in reducing the incidence of ARDS in individuals with severe sepsis (a condition characterized by an inflammatory response by the immune system throughout the whole body caused by infection) who are at high risk for the development of ARDS. All study participants will be randomized to receive placebo, bevacizumab 5 mg/kg or bevacizumab 10 mg/kg as a single intravenous dose in a double-blinded fashion in addition to traditional sepsis treatment.

ELIGIBILITY:
Inclusion Criteria:

* Clinical Diagnosis of Sepsis based on Modified Inflammatory Response Syndrome (SIRS) Criteria
* Evidence of a systemic response to infection
* 1 or more sepsis-induced organ failures modified from those as defined by Bernard, et al. (eg. PROWESS rhAPC study, NEJM)

Exclusion Criteria:

* Pregnant females
* Systolic blood pressure >170
* Diastolic blood pressure >110
* Preexisting proteinuria >0.3 g/24hr
* Known hypersensitivity to bevacizumab
* Subject or health care agent unable to provide written informed consent
* Diagnosis of lung cancer with active hemoptysis
* Patient not expected to survive 28 days independently of the septic episode due to severe underlying disease
* Presence of an advanced directive to withhold life-sustaining treatment
* Participation in another investigational study within 30 days of enrollment
* GI tract perforation and/or repair unless surgical incision is fully healed
* Any major surgery in the 28 days prior to enrollment
* Need for non-elective major surgery within 28 days
* Presence of enterocutaneous fistula (an abnormal connection between body cavities, in this case, from the intestine to the skin. Possible complication of surgery, where passageway progresses from intestine to surgery site to skin)
* Known or suspected tracheoesophageal fistula (an abnormal connection between the esophagus and the trachea)
* Current ICU stay of > 2 months prior to enrollment
* Need for therapeutic anti-coagulation

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-07; Primary Completion 2015-11 (Estimated); Study Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
Proportion of individuals progressing to meet RDS criteria as defined by the American- European ARDS consensus conference and as used by ARDSnet. | Day 28

SECONDARY OUTCOMES:
Ventilator-free days to Day 28 | Day 28
28 day all-cause mortality | Day 28
Proportion of subjects progressing to acute lung injury (who do not meet the definition at randomization) | Day 28
Worst PaO2/FiO2 ratio recorded following enrollment | Day 3 and 28
Change in PaO2/FiO2 ratio between Day 0 to Day 3 | Day 0 and Day 3
Change from baseline in number of non-lung organ failures using the Multi-Organ Dysfunction (MOD) score and Sepsis Organ Failure Assessment (SOFA) score | Day 0, Day 28
Proportion of subjects surviving to hospital discharge | Hospital Discharge Day
Vasopressor-free days | Day 28
Reversal of shock if present at randomization. | Day 28

CONTACTS AND LOCATIONS:
Overall Officials: Robert Kaner, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College-New York Presbyterian Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ware LB, Matthay MA. The acute respiratory distress syndrome. N Engl J Med. 2000 May 4;342(18):1334-49. doi: 10.1056/NEJM200005043421806. No abstract available. PMID 10793167
- [Background] Phua J, Badia JR, Adhikari NK, Friedrich JO, Fowler RA, Singh JM, Scales DC, Stather DR, Li A, Jones A, Gattas DJ, Hallett D, Tomlinson G, Stewart TE, Ferguson ND. Has mortality from acute respiratory distress syndrome decreased over time?: A systematic review. Am J Respir Crit Care Med. 2009 Feb 1;179(3):220-7. doi: 10.1164/rccm.200805-722OC. Epub 2008 Nov 14. PMID 19011152
- [Background] Kaner RJ, Ladetto JV, Singh R, Fukuda N, Matthay MA, Crystal RG. Lung overexpression of the vascular endothelial growth factor gene induces pulmonary edema. Am J Respir Cell Mol Biol. 2000 Jun;22(6):657-64. doi: 10.1165/ajrcmb.22.6.3779. PMID 10837361
- [Background] Rubenfeld GD, Caldwell E, Peabody E, Weaver J, Martin DP, Neff M, Stern EJ, Hudson LD. Incidence and outcomes of acute lung injury. N Engl J Med. 2005 Oct 20;353(16):1685-93. doi: 10.1056/NEJMoa050333. PMID 16236739
- [Background] National Heart, Lung, and Blood Institute Acute Respiratory Distress Syndrome (ARDS) Clinical Trials Network; Wiedemann HP, Wheeler AP, Bernard GR, Thompson BT, Hayden D, deBoisblanc B, Connors AF Jr, Hite RD, Harabin AL. Comparison of two fluid-management strategies in acute lung injury. N Engl J Med. 2006 Jun 15;354(24):2564-75. doi: 10.1056/NEJMoa062200. Epub 2006 May 21. PMID 16714767
- [Background] Kaner RJ, Crystal RG. Compartmentalization of vascular endothelial growth factor to the epithelial surface of the human lung. Mol Med. 2001 Apr;7(4):240-6. PMID 11471568
- [Background] Kaner RJ, Crystal RG. Pathogenesis of high altitude pulmonary edema: does alveolar epithelial lining fluid vascular endothelial growth factor exacerbate capillary leak? High Alt Med Biol. 2004 Winter;5(4):399-409. doi: 10.1089/ham.2004.5.399. PMID 15671629
- [Background] Hao Q, Wang L, Tang H. Vascular endothelial growth factor induces protein kinase D-dependent production of proinflammatory cytokines in endothelial cells. Am J Physiol Cell Physiol. 2009 Apr;296(4):C821-7. doi: 10.1152/ajpcell.00504.2008. Epub 2009 Jan 28. PMID 19176759
- [Background] Yano K, Liaw PC, Mullington JM, Shih SC, Okada H, Bodyak N, Kang PM, Toltl L, Belikoff B, Buras J, Simms BT, Mizgerd JP, Carmeliet P, Karumanchi SA, Aird WC. Vascular endothelial growth factor is an important determinant of sepsis morbidity and mortality. J Exp Med. 2006 Jun 12;203(6):1447-58. doi: 10.1084/jem.20060375. Epub 2006 May 15. PMID 16702604
- [Background] van der Flier M, van Leeuwen HJ, van Kessel KP, Kimpen JL, Hoepelman AI, Geelen SP. Plasma vascular endothelial growth factor in severe sepsis. Shock. 2005 Jan;23(1):35-8. doi: 10.1097/01.shk.0000150728.91155.41. PMID 15614129
- [Background] Tsao PN, Chan FT, Wei SC, Hsieh WS, Chou HC, Su YN, Chen CY, Hsu WM, Hsieh FJ, Hsu SM. Soluble vascular endothelial growth factor receptor-1 protects mice in sepsis. Crit Care Med. 2007 Aug;35(8):1955-60. doi: 10.1097/01.CCM.0000275273.56547.B8. PMID 17568329
- [Background] Watanabe M, Boyer JL, Crystal RG. Genetic delivery of bevacizumab to suppress vascular endothelial growth factor-induced high-permeability pulmonary edema. Hum Gene Ther. 2009 Jun;20(6):598-610. doi: 10.1089/hum.2008.169. PMID 19254174
- [Background] Pepe PE, Potkin RT, Reus DH, Hudson LD, Carrico CJ. Clinical predictors of the adult respiratory distress syndrome. Am J Surg. 1982 Jul;144(1):124-30. doi: 10.1016/0002-9610(82)90612-2. PMID 7091520
- [Background] Bernard GR, Artigas A, Brigham KL, Carlet J, Falke K, Hudson L, Lamy M, Legall JR, Morris A, Spragg R. The American-European Consensus Conference on ARDS. Definitions, mechanisms, relevant outcomes, and clinical trial coordination. Am J Respir Crit Care Med. 1994 Mar;149(3 Pt 1):818-24. doi: 10.1164/ajrccm.149.3.7509706.
- [Background] Nolan A, Weiden MD, Thurston G, Gold JA. Vascular endothelial growth factor blockade reduces plasma cytokines in a murine model of polymicrobial sepsis. Inflammation. 2004 Oct;28(5):271-8. doi: 10.1007/s10753-004-6050-3. PMID 16134000
- [Background] Wakelee H. Antibodies to vascular endothelial growth factor in non-small cell lung cancer. J Thorac Oncol. 2008 Jun;3(6 Suppl 2):S113-8. doi: 10.1097/JTO.0b013e318174e993. PMID 18520292
- [Background] Watanabe M, Boyer JL, Hackett NR, Qiu J, Crystal RG. Genetic delivery of the murine equivalent of bevacizumab (avastin), an anti-vascular endothelial growth factor monoclonal antibody, to suppress growth of human tumors in immunodeficient mice. Hum Gene Ther. 2008 Mar;19(3):300-10. doi: 10.1089/hum.2007.109. PMID 18324912
- [Background] Shapiro NI, Yano K, Okada H, Fischer C, Howell M, Spokes KC, Ngo L, Angus DC, Aird WC. A prospective, observational study of soluble FLT-1 and vascular endothelial growth factor in sepsis. Shock. 2008 Apr;29(4):452-7. doi: 10.1097/shk.0b013e31815072c1. PMID 18598002